CLINICAL TRIAL: NCT01381731
Title: A Double-masked, Randomized, Placebo-controlled,Pilot Study of Diquafosol Tetrasodium in Subjects Following Photorefractive Keratectomy (PRK)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 03-201
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Photorefractive Keratectomy
Keywords: post PRK wound healing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Diquafosol tetrasodium ophthalmic solution 2% (Experimental): topical ophthalmic solution
  Interventions: Drug: diquafosol tetrasodium ophthalmic solution 2%
- Placebo (Placebo Comparator): saline ophthalmic solution
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: diquafosol tetrasodium ophthalmic solution 2% — opthalmic solution 2 drops in each eye QID
  Arms: Diquafosol tetrasodium ophthalmic solution 2%
Drug: placebo — opthalmic solution 2 drops in each eye QID
  Arms: Placebo

SUMMARY:
The objectives of this trial are to:

* Assess the safety and tolerability of diquafosol tetrasodium ophthalmic solution versus placebo following one week of treatment in subjects undergoing photorefractive keratectomy (PRK).
* Evaluate the potential of diquafosol to accelerate corneal wound healing/re-epithelialization following PRK.

ELIGIBILITY:
Inclusion Criteria:

* between age 18 - 45 years old
* candidate for bilateral PRK

Exclusion Criteria:

* dry eye disease
* any corneal pathologies
* previous corneal or intraocular surgeries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2005-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Healing time | 12 weeks

SECONDARY OUTCOMES:
Adverse events | 12 weeks